CLINICAL TRIAL: NCT01123343
Title: CLINICAL EVALUATION OF THE TRUEVISION 3D VISUALIZATION AND GUIDANCE SYSTEM FOR MICROSURGERY: LRI AND CAPSULORHEXIS TEMPLATES
Brief Title: Clinical Evaluation of TrueVision System: LRI and Capsulorhexis Templates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TrueVision Systems, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVS-2009-001
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Subjects Undergoing Cataract Surgery and Insertion of IOL
Keywords: limbal relaxing incision; LRI; capsulorhexis; surgical guidance; 3d visualization
MeSH Terms: interventions — Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LRI Templates (Active Comparator): To evaluate the ability of the TRUEVISION 3D VISUALIZATION AND GUIDANCE SYSTEM FOR MICROSURGERY to provide the ophthalmic surgeon appropriate alignment, orientation and sizing information during cataract or refractive lens exchange surgery compared to the current standard of care (manual markings or heuristic techniques) for LRI.
  Interventions: Device: TrueVision 3D Visualization and Guidance System for MicroSurgery
- Capsulorhexis Templates (Active Comparator): To evaluate the ability of the TRUEVISION 3D VISUALIZATION AND GUIDANCE SYSTEM FOR MICROSURGERY to provide the ophthalmic surgeon appropriate alignment, orientation and sizing information during cataract or refractive lens exchange surgery compared to the current standard of care (manual markings or heuristic techniques) for Capsulorhexis.
  Interventions: Device: TrueVision 3D Visualization and Guidance System for MicroSurgery

INTERVENTIONS:
Device: TrueVision 3D Visualization and Guidance System for MicroSurgery — Adjunct imaging tool (to the microscope oculars) that provides onscreen video guidance for alignment, orientation, and sizing during eye surgery, based on a surgeon's defined nomogram

SUMMARY:
To evaluate the ability of the TRUEVISION 3D VISUALIZATION AND GUIDANCE SYSTEM FOR MICROSURGERY to provide the ophthalmic surgeon appropriate alignment, orientation and sizing information during cataract or refractive lens exchange surgery. Device images, safety results and surgeon questionnaire will demonstrate that the TrueVision system provides clear images to assist surgeons during LRI or capsulorhexis procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eye with no previous ocular surgery
* Natural lens for which phacoemulsification extraction and posterior IOL implantation is planned
* Clear intraocular media other than cataract
* Potential visual acuity 20/30 or better
* Able to comply with preop and postop examination procedures
* Signed and dated informed consent

Exclusion Criteria:

* Keratometric astigmatism > 2.5 diopters
* Corneal pathology potentially affecting topography including corneal degeneration
* Irregular astigmatism
* Macular degeneration or any other macular disease which reduces potential acuity
* Previous corneal surgery (including LASIK, radial keratotomy, penetrating keratoplasty, etc)
* Use of systemic or ocular medications that affects vision
* Acute or chronic systemic or ocular disease or illness that would increase risk or confound study results
* Use of Flomax or any other medication which negatively impacts surgical outcomes
* History of ocular trauma or ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the TrueVision system provides clear images to assist during LRI or capsulorhexis procedures | one month

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, Study Director — Oregon Eye Associates; Robert Weinstock, MD, Principal Investigator — Eye Institute of West Florida; Jason Stahl, MD, Principal Investigator — Durrie Vision; Douglas Katsev, MD, Principal Investigator — Sansum Clinic
Locations (1):
- Drs. Fine, Hoffman and Packer, Eugene, Oregon, United States